CLINICAL TRIAL: NCT06035484
Title: Effect of Seat Height and Angle on Wheelchair Foot Propulsion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Ed Giesbrecht, Associate professor, University of Manitoba
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HS25835 (H2023:027)
Record Dates: First submitted 2023-02-07; First posted 2023-09-13 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Healthy
Keywords: Manual Wheelchair; Bilateral propulsion; Foot propulsion

STUDY DESIGN:
Intervention Model Description: Within-subjects repeated measures design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- LL & 0 (Experimental): Wheelchair seat height will be positioned at lower leg length and set inclination will be zero
  Interventions: Other: Seat height; Other: Seat inclination
- LL + 1 (Experimental): Wheelchair seat height will be positioned at the participant's leg length plus one inch with an inclination of zero
  Interventions: Other: Seat height
- LL - 1 (Experimental): Wheelchair seat height will be positioned at the participant's leg length minus one inch with an inclination of zero
  Interventions: Other: Seat height
- LL - 2 (Experimental): Wheelchair seat height will be positioned at the participant's leg length minus two inches with an inclination of zero
  Interventions: Other: Seat height
- LL - 3 (Experimental): Wheelchair seat height will be positioned at the participant's leg length minus three inches with an inclination of zero
  Interventions: Other: Seat height
- 3 degrees Inclination (Experimental): Wheelchair seat height will be positioned at the participant's leg length with a forward seat inclination of 3 degrees
  Interventions: Other: Seat inclination
- 6 degrees Inclination (Experimental): Wheelchair seat height will be positioned at the participant's leg length with a forward seat inclination of 6 degrees
  Interventions: Other: Seat inclination
- 9 degrees Inclination (Experimental): Wheelchair seat height will be positioned at the participant's leg length with a forward seat inclination of 9 degrees
  Interventions: Other: Seat inclination

INTERVENTIONS:
Other: Seat height — Seat height of a manual wheelchair will be changed according the different arms specified. The participant will complete a course in the manual wheelchair with each arm.
  Arms: LL & 0; LL + 1; LL - 1; LL - 2; LL - 3
Other: Seat inclination — Seat inclination of a manual wheelchair will be changed according the different arms specified. The participant will complete a course in the manual wheelchair with each arm.
  Arms: 3 degrees Inclination; 6 degrees Inclination; 9 degrees Inclination; LL & 0

SUMMARY:
The purpose of the project is to explore the effect of differences in seat height and seat angle on bilateral foot propulsion using a manual wheelchair. The objectives of the study are to determine whether differences in seat height and seat angle impact: a) propulsion speed; b) knee range of motion used during propulsion; c) effectiveness of foot propulsion gait; and d) perceived difficulty with foot propulsion.

A repeated measures designs allows comparison between 5 different seat height conditions and 4 different seat angle conditions to determine whether there are significant differences in outcome, and if so, which conditions provide better outcomes. Participants will propel a customized MWC through a standardized course using each seat configuration; the sequence will be randomized to reduce any learning effects.

ELIGIBILITY:
Inclusion Criteria:

* student in College of Rehabilitation Sciences enrolled in Master of Occupational Therapy, Master of Physical Therapy, or Bachelor of Respiratory Therapy program at the University of Manitoba.
* Able-bodied individuals

Exclusion Criteria:

* Students whose hip width exceeds 21 inches or lower leg length is shorter than 16 inches will be excluded as the test manual wheelchair will not accommodate these dimensions.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2023-04-20 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Propulsion speed | ~30-60 seconds
  Speed will be determined via video recording. Two outcomes will be determined initial 10m and total test course
Knee range of motion | ~30-60 seconds
  Xsens sensors and mobile app will be used to determine the positions of the thigh and lower leg and knee joint angle will be obtained from the difference between these positions.
Effectiveness of foot propulsion gait | ~30-60 seconds
  Evaluated using the Wheelchair Propulsion Test developed by Askari et al. (2013). Simple, valid and reliable measure of propulsion for either upper or lower extremity propulsion techniques.
Perceived difficulty with foot propulsion | ~30-60 seconds
  Participant will provide subjective evaluations of how difficult they found foot propulsion after each trial, using Perceived Difficulty Questionnaire (Heinrichs et al., 2021).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No
Data will not be shared outside of the principle and student investigator's conducting this study.

REFERENCES:
- [Background] Askari S, Kirby RL, Parker K, Thompson K, O'Neill J. Wheelchair propulsion test: development and measurement properties of a new test for manual wheelchair users. Arch Phys Med Rehabil. 2013 Sep;94(9):1690-8. doi: 10.1016/j.apmr.2013.03.002. Epub 2013 Mar 14. PMID 23499781
- [Background] Heinrichs ND, Kirby RL, Smith C, Russell KFJ, Theriault CJ, Doucette SP. Effect of seat height on manual wheelchair foot propulsion, a repeated-measures crossover study: part 1 - wheeling forward on a smooth level surface. Disabil Rehabil Assist Technol. 2021 Nov;16(8):831-839. doi: 10.1080/17483107.2020.1741036. Epub 2020 Apr 2. PMID 32238086